CLINICAL TRIAL: NCT02703350
Title: Pharmacokinetics, Glucodynamics, Safety, and Tolerability of LY900014 in Patients With Type 1 Diabetes Mellitus on Multiple Daily Insulin Injection Therapy
Brief Title: A Study of LY900014 in Participants With Type 1 Diabetes on Insulin Injection Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16068; I8B-FW-ITRG (Other: Eli Lilly and Company); 2015-004737-27 (EudraCT Number)
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY900014 - Test (Part A) (Experimental): Individualized doses of LY900014 administered by injection under the skin once in each of 3 periods
  Interventions: Drug: LY900014
- Insulin Lispro - Reference (Part A) (Active Comparator): Individualized doses of insulin lispro reference formulation administered by injection under the skin once in each of 3 periods
  Interventions: Drug: Insulin Lispro
- LY900014 - Test (Part B) (Experimental): Individualized doses of LY900014 administered by injection under the skin immediately before each meal for 14 days
  Interventions: Drug: LY900014
- Insulin Lispro - Reference (Part B) (Active Comparator): Individualized doses of insulin lispro reference formulation administered by injection under the skin immediately before each meal for 14 days
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY900014 — Administered subcutaneously (SC)
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014 - Test (Part A); LY900014 - Test (Part B)
Drug: Insulin Lispro — Administered SC
  Other Names: LY275585
  Arms: Insulin Lispro - Reference (Part A); Insulin Lispro - Reference (Part B)

SUMMARY:
The study will be conducted in participants with type1 diabetes on insulin injection therapy to investigate how the body processes LY900014 and the effect of LY900014 on blood sugar levels. Side effects and tolerability will be documented. The study will be conducted in two parts (Part A and Part B) to achieve its objectives. Participants are expected to enroll in both parts.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female participants with Type 1 Diabetes Mellitus (T1DM) on a stable multiple daily injection regimen with a short-acting as well as a long-acting insulin
* Have a body mass index (BMI) ranging from 18.5 to 33.0 kilogram per square meter (kg/m²), inclusive, at screening
* Have blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results acceptable for the study
* Have had no episodes of severe hypoglycemia in the past 6 months (requiring assistance in treatment by a second party)
* Have venous access sufficient to allow for blood sampling
* Have provided written consent and are willing to follow study procedures and commit to the study duration

Exclusion Criteria:

* Are currently enrolled, or have participated within the last 30 days, in a clinical trial or any other type of medical research judged to be incompatible with this study
* Have previously completed or withdrawn from this study
* Have or used to have health problems that, in the opinion of the doctor, could make it unsafe to participate in the study
* Had blood loss of more than 500 milliliters (mL) within the last month
* Are treated with a continuous subcutaneous insulin infusion (insulin pump)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Mainz, Germany

REFERENCES:
- See also: Click here for more information about this study: A Study of LY900014 in Participants With Type 1 Diabetes on Insulin Injection Therapy — http://www.lillytrialguide.com/EN-US/studies/diabetes/itrg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two-part study compared individualized doses of LY900014 (Test) to insulin lispro (Reference). Part A: LY900014 or insulin lispro once subcutaneously (SC) before, at, or after start of meal in each of 6 periods. Minimum 1 day washout. Part B: LY900014 or insulin lispro SC before meals for 14 days. Participants were expected to complete both parts.
Groups:
- Part A Sequence 1, ABFCED: A = LY900014 Test (15 minutes [mins] before meal). B = LY900014 Test (at mealtime). C = LY900014 Test (15 mins after start of meal). D = Insulin Lispro Reference (15 mins before meal). E = Insulin Lispro Reference (at mealtime). F = Insulin Lispro Reference (15 mins after start of meal).
- Part A Sequence 2, BCADFE; Part A Sequence 3, CDBEAF; Part A Sequence 4, DECFBA; Part A Sequence 5, EFDACB; Part A Sequence 6, FAEBDC: A = LY900014 Test (15 mins before meal). B = LY900014 Test (at mealtime). C = LY900014 Test (15 mins after start of meal). D = Insulin Lispro Reference (15 mins before meal). E = Insulin Lispro Reference (at mealtime). F = Insulin Lispro Reference (15 mins after start of meal).
- Part B LY900014 (Test): Individualized doses of LY900014 Test administered SC immediately before meals for 14 days.
- Part B Insulin Lispro (Reference): Individualized doses of Insulin Lispro Reference administered SC immediately before meals for 14 days.
Period: Period One (Part A)
Arm/Group | Part A Sequence 1, ABFCED | Part A Sequence 2, BCADFE | Part A Sequence 3, CDBEAF | Part A Sequence 4, DECFBA | Part A Sequence 5, EFDACB | Part A Sequence 6, FAEBDC | Part B LY900014 (Test) | Part B Insulin Lispro (Reference)
Started | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Received Study Drug | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period Two (Part A)
Arm/Group | Part A Sequence 1, ABFCED | Part A Sequence 2, BCADFE | Part A Sequence 3, CDBEAF | Part A Sequence 4, DECFBA | Part A Sequence 5, EFDACB | Part A Sequence 6, FAEBDC | Part B LY900014 (Test) | Part B Insulin Lispro (Reference)
Started | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Received Study Drug | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period Three (Part A)
Arm/Group | Part A Sequence 1, ABFCED | Part A Sequence 2, BCADFE | Part A Sequence 3, CDBEAF | Part A Sequence 4, DECFBA | Part A Sequence 5, EFDACB | Part A Sequence 6, FAEBDC | Part B LY900014 (Test) | Part B Insulin Lispro (Reference)
Started | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Received Study Drug | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period Four (Part A)
Arm/Group | Part A Sequence 1, ABFCED | Part A Sequence 2, BCADFE | Part A Sequence 3, CDBEAF | Part A Sequence 4, DECFBA | Part A Sequence 5, EFDACB | Part A Sequence 6, FAEBDC | Part B LY900014 (Test) | Part B Insulin Lispro (Reference)
Started | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Received Study Drug | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period Five (Part A)
Arm/Group | Part A Sequence 1, ABFCED | Part A Sequence 2, BCADFE | Part A Sequence 3, CDBEAF | Part A Sequence 4, DECFBA | Part A Sequence 5, EFDACB | Part A Sequence 6, FAEBDC | Part B LY900014 (Test) | Part B Insulin Lispro (Reference)
Started | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Received Study Drug | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period Six (Part A)
Arm/Group | Part A Sequence 1, ABFCED | Part A Sequence 2, BCADFE | Part A Sequence 3, CDBEAF | Part A Sequence 4, DECFBA | Part A Sequence 5, EFDACB | Part A Sequence 6, FAEBDC | Part B LY900014 (Test) | Part B Insulin Lispro (Reference)
Started | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Received Study Drug | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A Sequence 1, ABFCED | Part A Sequence 2, BCADFE | Part A Sequence 3, CDBEAF | Part A Sequence 4, DECFBA | Part A Sequence 5, EFDACB | Part A Sequence 6, FAEBDC | Part B LY900014 (Test) | Part B Insulin Lispro (Reference)
Started (Participants who completed all six periods in Part A were eligible for Part B.) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15
Received Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants: Individualized doses of LY900014 (Test) or insulin lispro (Reference) administered once SC at various mealtime intervals in each of six periods (Part A) and immediately before meals for 14 days (Part B).
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 30

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under the Concentration Curve From Time Zero to 5 Hours (AUC[0-5h]) (Part A)
Description: PK: Insulin Lispro AUC(0-5h) (Part A)
Time Frame: Day 1: 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150,180, 240, 300 minutes post dose for each treatment
Population: All participants in Part A who received study drug and had evaluable PK data. For one participant in the LY900014 - Test (Part A) group, the insulin lispro PK profile (period three) was excluded from the mean PK analysis, as there was no absorption phase observed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole*hour per liter (pmol*h/L)
Groups:
- Insulin Lispro - Reference (Part A): Individualized doses of insulin lispro (Reference) administered once SC in three of six periods.
- LY900014 - Test (Part A): Individualized doses of LY900014 (Test) administered once SC in three of six periods.
Arm/Group | Insulin Lispro - Reference (Part A) | LY900014 - Test (Part A)
Number analyzed (Participants) | 30 | 30
picomole*hour per liter (pmol*h/L) | 719 (52) | 783 (51)

2. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under the Concentration Curve From Time Zero to 5 Hours (AUC[0-5h]) (Part B)
Description: PK: Insulin Lispro AUC(0-5h) (Part B)
Time Frame: Days 1 and 14: 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150,180, 240, 300 minutes post dose for each treatment
Population: All participants in Part B who received study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol*h/L
Groups:
- Insulin Lispro - Reference (Part B): Individualized doses of insulin lispro (Reference) administered SC immediately before each meal for 14 days.
- LY900014 - Test (Part B): Individualized doses of LY900014 (Test) administered SC immediately before each meal for 14 days.
Arm/Group | Insulin Lispro - Reference (Part B) | LY900014 - Test (Part B)
Number analyzed (Participants) | 15 | 15
pmol*h/L
  Day 1 | 751 (40) | 780 (63)
  Day 14 | 718 (50) | 771 (61)

3. Secondary Outcome: Pharmacodynamics (PD): Area Under the Concentration Curve From Time Zero to 5 Hours (AUC[0-5h]) of Glucose Relative to a Mixed Meal Tolerance Test (MMTT) (Part A)
Description: PD: AUC(0-5h) of Glucose Relative to a MMTT (Part A)
Time Frame: Day 1: -30, -15, 0, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120, 135, 150, 165, 180, 195, 210, 225, 240, 300 minutes
Population: All participants in Part A who received study drug immediately before a meal (0 min) and had evaluable PD data. Data were excluded if the participant did not keep identical insulin lispro dose during the MMTT assessments, did not complete the entire test meal, or had significant changes in nutrient consumption of the test meal.
Measure: Mean (Standard Deviation); unit: milligram*hour/deciliter (mg*h/dL)
Groups:
- Insulin Lispro - Reference 0 Min (Part A): Individualized doses of insulin lispro (Reference) administered once SC immediately before meal in one of six periods.
- LY900014 - Test 0 Min (Part A): Individualized doses of LY900014 (Test) administered once SC immediately before meal in one of six periods.
Arm/Group | Insulin Lispro - Reference 0 Min (Part A) | LY900014 - Test 0 Min (Part A)
Number analyzed (Participants) | 29 | 27
milligram*hour/deciliter (mg*h/dL) | 495 (161) | 537 (184)

4. Secondary Outcome: Pharmacodynamics (PD): Area Under the Concentration Curve From Time Zero to 5 Hours (AUC[0-5h]) of Glucose Relative to a Mixed Meal Tolerance Test (MMTT) (Part B)
Description: PD: AUC(0-5h) of Glucose Relative to a MMTT (Part B)
Time Frame: Days 1 and 14: Day 1: -30, -15, 0, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120, 135, 150, 165, 180, 195, 210, 225, 240, 300 minutes in each study period
Population: All participants in Part B who received study drug and had evaluable PD data. Data were excluded if the participant did not keep identical insulin lispro dose during the MMTT assessments, did not complete the entire test meal, or had significant changes in nutrient consumption of the test meal.
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Insulin Lispro - Reference (Part B) | LY900014 - Test (Part B)
Number analyzed (Participants) | 15 | 14
mg*h/dL
  Day 1: number analyzed (Participants) | 13 | 14
  Day 1 | 533 (205) | 404 (131)
  Day 14 | 547 (239) | 411 (130)

ADVERSE EVENTS:
Groups:
- Insulin Lispro - Reference -15 Min (Part A): Individualized doses of insulin lispro (Reference) administered once SC 15 minutes prior to meal in one of six periods.
- Insulin Lispro - Reference +15 Min (Part A): Individualized doses of insulin lispro (Reference) administered once SC 15 minutes after start of meal in one of six periods.
- LY900014 - Test -15 Min (Part A): Individualized doses of LY900014 (Test) administered once SC 15 minutes prior to meal in one of six periods.
- LY900014 - Test +15 Min (Part A): Individualized doses of LY900014 (Test) administered once SC 15 minutes after start of meal in one of six periods.
- Insulin Lispro Open Label - (Part A): Individualized doses of insulin lispro administered SC between periods.
- Insulin Lispro - Reference (Part B): Individualized doses of insulin lispro (Reference) administered SC immediately before meals for 14 days.
- LY900014 - Test (Part B): Individualized doses of LY900014 (Test) administered SC immediately before meals for 14 days.
- Insulin Lispro Open Label - (Part B): Individualized doses of insulin lispro administered SC immediately before meals.
Arm/Group | Insulin Lispro - Reference -15 Min (Part A) | Insulin Lispro - Reference 0 Min (Part A) | Insulin Lispro - Reference +15 Min (Part A) | LY900014 - Test -15 Min (Part A) | LY900014 - Test 0 Min (Part A) | LY900014 - Test +15 Min (Part A) | Insulin Lispro Open Label - (Part A) | Insulin Lispro - Reference (Part B) | LY900014 - Test (Part B) | Insulin Lispro Open Label - (Part B)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/15 | 0/15 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 1/30 | 0/30 | 0/30 | 0/30 | 1/30 | 0/30 | 2/15 | 1/15 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro - Reference -15 Min (Part A) (N=30) | Insulin Lispro - Reference 0 Min (Part A) (N=30) | Insulin Lispro - Reference +15 Min (Part A) (N=30) | LY900014 - Test -15 Min (Part A) (N=30) | LY900014 - Test 0 Min (Part A) (N=30) | LY900014 - Test +15 Min (Part A) (N=30) | Insulin Lispro Open Label - (Part A) (N=30) | Insulin Lispro - Reference (Part B) (N=15) | LY900014 - Test (Part B) (N=15) | Insulin Lispro Open Label - (Part B) (N=30)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days